CLINICAL TRIAL: NCT01103375
Title: A Phase I Single Arm Open Label Study of Erlotinib and 13-cis-Retinoic Acid (CRA) in Patients With Recurrent Malignant Gliomas
Brief Title: Erlotinib Hydrochloride and Isotretinoin in Treating Patients With Recurrent Malignant Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012306; NCI-2010-00132 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 91209 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Oligodendroglioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzyme inhibitor, immunotherapy) (Experimental): Patients receive isotretinoin PO QD on days 1-21 and erlotinib hydrochloride PO QD on days 1-28.
  Interventions: Drug: erlotinib hydrochloride; Drug: isotretinoin; Other: laboratory biomarker analysis; Genetic: protein expression analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: isotretinoin — Given PO
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret
Other: laboratory biomarker analysis — Correlative study
Genetic: protein expression analysis — Correlative study

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib hydrochloride when given with isotretinoin in treating patients with recurrent malignant glioma. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Isotretinoin may help cells that are involved in the body's immune response to work better. Giving erlotinib hydrochloride together with isotretinoin may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II doses of erlotinib (erlotinib hydrochloride) and 13-cis-retinoic acid (CRA) when administered to adults with recurrent malignant glioma who are not receiving cytochrome P450 enzyme-inducing antiepileptic drugs (EIAEDs).

SECONDARY OBJECTIVES:

I. To assess dose-related toxicities. II. To measure 6 month progression-free survival and overall survival. III. To estimate response rates in those patients with measurable disease. IV. To evaluate for epidermal growth factor receptor (EGFR)vIII, phosphatase and tensin homolog (PTEN), cyclin D1, cyclin E, and RARbeta1 expression in tumor samples from enrolled patients as predictors of clinical benefit from this combination.

OUTLINE: This is a dose-escalation study.

Patients receive isotretinoin orally (PO) once daily (QD) on days 1-21 and erlotinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven malignant glioma (glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendroglioma, or anaplastic mixed oligoastrocytoma) which is progressive or recurrent after radiation therapy +/- chemotherapy; patients with previous low grade glioma who progressed after radiotherapy +/- chemotherapy and are biopsied and found to have a high grade glioma are eligible Karnofsky performance status of >= 60% Patients - both males and females - with reproductive potential (i.e., premenopausal or menopausal for less than 1 year and not surgically sterilized) must practice at least 2 contraceptive measures throughout the study Patients must be registered and meet all the requirements of iPLEDGE in order to receive 13-cis-Retinoic Acid (CRA) Patients must provide verbal and written informed consent to participate in the study Patients must have a Mini Mental Status Exam score >= 15 Patients must have a 12-lead electrocardiogram (EKG) without evidence of any clinically significant abnormalities Absolute neutrophil count (ANC) >= 1,500/mm^3 Platelets >= 100,000/mm^3 Aspartate aminotransferase (AST) =< 2.5 upper limit of normal (ULN) (ULN = 50 U/L) Alanine aminotransferase (ALT) =< 2.5 ULN (ULN = 50 U/L) Total Bilirubin =< 1.5 mg/dL Alkaline phosphatase (Alk. Phos) =< 5X ULN (ULN = 125 U/dL) Estimated (Estim.) creatinine (Cr) Clearance > 50 ml/min Fasting total cholesterol < 300 mg/dL Fasting triglycerides < 250 mg/dL Two separate, laboratory pregnancy tests within 14 days of registration (for women of childbearing potential) Patients must have recovered from the toxicity of prior therapy; specifically, there must be at least a 3 month interval from the completion of the most recent course of radiation therapy, at least a 3 month interval from the implantation of Gliadel wafer(s), at least a 3 week interval from the completion of a non-nitrosourea-containing chemotherapy regimen, and at least a 6 week interval from the completion of a nitrosourea-containing chemo-regimen

Exclusion Criteria:

Pregnant or breast-feeding women Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, severe cardiovascular disease including recent (< 6 months) myocardial infarction, severe psychiatric illness that would limit compliance with study requirements, or any other disorder that would be incompatible with the study therapy Any history of inflammatory bowel disease Any history of uncontrolled depression, any history of hospitalization for depression, or any history of suicidal thoughts or attempt(s) Patients receiving concurrent therapy for their tumor (with the exception of steroids) Must have at least a 10 day interval from last dose of vitamin A, tetracyclines, micro-dosed progesterone preparations, norethindrone/ethinyl estradiol, St. John's Wort, fish oil supplements, or phenytoin or other P450 enzyme inducing antiepileptic drugs Current smokers (Smoking >= 11 cigarettes per day), as smoking increases metabolism and decreases serum levels of erlotinib Participants may not have received prior EGFR inhibitors for any disease Patients with a history of allergic reactions to 13-cis-retinoic acid (CRA) or compounds of similar biologic or chemical composition to CRA Known allergy to proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Recommended phase II doses of erlotinib hydrochloride and isotretinoin | 3 weeks
  At least 3 patients will be treated at each dose level and the maximum tolerated dose (MTD) will be determined. Patients will be evaluated for dose-limiting toxicity (DLT) in the first 3 weeks on protocol.

SECONDARY OUTCOMES:
Toxicity as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 | Up to 2 years
Progression-free survival | At 6 months
Overall survival | At 6 months
Response rates (complete or partial response) | Up to 2 years
EGFRvIII, PTEN, cyclin D1, cyclin E, and RARbeta1 expression in tumor samples | Pre-study

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States